CLINICAL TRIAL: NCT00873912
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of a New 6:2 Influenza Virus Reassortant in Healthy Adults
Brief Title: A Prospective Study to Evaluate the Safety of a New Monovalent Intranasal Influenza Vaccine
Acronym: MI-MA205
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Elissa Malkin, DO/Dir Clinical Development, MedImmune, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-MA205
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: influenza; FluMist
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monovalent influenza virus vaccine (Experimental): Frozen monovalent vaccine containing new strain
  Interventions: Biological: Monovalent influenza virus vaccine
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Monovalent influenza virus vaccine — Monovalent vaccine was supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose-phosphate buffer, egg allantoic fluid, and approximately 10^7 FFU (fluorescent focus units) of the cold-adapted, attenuated, 6:2 reassortant influenza strain B/Brisbane/60/2008 (Victoria lineage).
  Arms: Monovalent influenza virus vaccine
Biological: Placebo — Placebo was supplied in intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer.
  Arms: Placebo

SUMMARY:
This prospective annual release study was designed to assess the safety of a monovalent influenza virus vaccine using a new strain recommended for the 2009-2010 influenza season not previously contained in the trivalent intranasal FluMist vaccine. Three hundred healthy adults received a single dose of vaccine or placebo and were followed for 180 days.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, placebo-controlled release study enrolled 300 healthy adults 18 to 49 years of age. Eligible participants were randomly assigned in a 4:1 fashion to receive a single dose of monovalent vaccine or placebo by intranasal spray. This study was conducted at multiple sites in the United States. Randomization was stratified by site.

Each participant received one dose of investigational product on Day 1. The duration of study participation for each participant was the time from receipt of investigational product through 180 days after receipt of investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 49 years of age (not yet reached their 50th birthday) at the time of investigational product administration
* Healthy by medical history and physical exam
* Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act [HIPAA] in the United States of America [USA], European Union [EU] Data Privacy Directive in the EU) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Females of childbearing potential, unless surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), had sterile male partner, were premenarchal or at least 2 years postmenopausal, or practiced abstinence, must have used 2 effective methods of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner) for at least 30 days prior to dosing with investigational product, and must have agreed to continue using such precautions for at least 90 days after dosing with investigational product; cessation of birth control after this point was to be discussed with a responsible physician. The subject must also have had a negative serum or urine pregnancy test within 14 days prior to investigational product administration (if screening and administration of investigational product did not occur on the same day) and on the day of investigational product administration prior to randomization
* Males, unless surgically sterile, must have used 2 effective methods of birth control with a female partner and must have agreed to continue using such contraceptive precautions for at least 30 days after dosing with investigational product (from Day 1 through Day 31 of the study)
* Subject available by telephone
* Ability to understand and comply with the requirements of the protocol, as judged by the investigator
* Ability to complete follow-up period of 180 days after dosing as required by the protocol

Exclusion Criteria:

* History of hypersensitivity to any component of the vaccine, including egg or egg protein or serious, life-threatening, or severe reactions to previous influenza vaccinations
* History of hypersensitivity to gentamicin
* Any condition for which the inactivated influenza vaccine was indicated, including chronic disorders of the pulmonary or cardiovascular systems (eg, asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (> 100.0°F oral or equivalent) and/or clinically significant respiratory illness (eg, cough or sore throat) within 14 days prior to randomization
* Any known immunosuppressive condition or immune deficiency disease, including human immunodeficiency virus [HIV] infection, or ongoing immunosuppressive therapy
* History of Guillain-Barré syndrome
* A household contact who was severely immunocompromised (eg, hematopoietic stem cell transplant recipient, during those periods in which the immunocompromised individual required care in a protective environment); subject should additionally have avoided close contact with severely immunocompromised individuals for at least 21 days after receipt of investigational product
* Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 30 days after the dose of investigational product (use of licensed agents for indications not listed in the package insert was permitted)
* Expected receipt of anti-pyretic or analgesic medication on a daily or every other day basis from randomization through 14 days after receipt of investigational product
* Administration of intranasal medications within 14 days prior to randomization, or expected receipt through 14 days after administration of investigational product
* Known or suspected mitochondrial encephalomyopathy
* Nursing mother
* Any condition (eg, chronic cough, allergic rhinitis) that, in the opinion of the investigator, would have interfered with evaluation of the investigational product or interpretation of subject safety or study results
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-05; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Malkin, D.O., Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Covance CRU, Inc., Daytona Beach, Florida
  - Covance CRU, Inc, Portland, Oregon
  - Covance CRU, Inc, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 300 subjects were randomized into the study between 26May2009 and 27May2009 at 3 sites in the USA.
Pre-assignment Details: Each site enrolled and randomized 80 subjects in the monovalent vaccine group and 20 subjects in the placebo group
Groups:
- Monovalent Influenza Virus Vaccine: Frozen monovalent vaccine containing the new strain was supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose-phosphate buffer, egg allantoic fluid, and approximately 10^7 fluorescent focus units (FFU) of influenza virus type B/Brisbane/60/2008 (Victoria lineage). A single dose of investigational product was administered on Day 1.
- Placebo: Placebo was supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose-phosphate buffer and egg allantoic fluid. A single dose of investigational product was administered on Day 1.
Period: Overall Study
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Started | 240 | 60
Completed | 237 | 60
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo | Total
Number analyzed (Participants) | 240 | 60 | 300
Age Continuous [Mean (Standard Deviation); unit: years] | 32.2 (8.1) | 30.9 (8.6) | 31.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 33 | 157
  Male | 116 | 27 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 10 | 46
  Not Hispanic or Latino | 204 | 50 | 254
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 7 | 2 | 9
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 5 | 23
  White | 206 | 50 | 256
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
  Other | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 240 | 60 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Fever, Defined as Oral Temperature ≥ 101°F
Description: The percentage of subjects with fever was compared between the two treatment groups based on the upper limit of the two-sided 95% exact confidence interval (CI) for the rate difference (monovalent vaccine minus placebo). The upper limit of the two-sided 95% CI was evaluated against the pre-specified equivalence criterion of 5 percentage points which corresponded to the following hypotheses: - H0 (null): rate difference ≥ 5 percentage points, - HA (alternative): rate difference < 5 percentage points.
Time Frame: Days 1-8 after vaccination
Population: The Safety Population includes all subjects who received at least one dose of investigational product and experienced any follow-up for safety. Treatment group was assigned based on the actual investigational product received.
Measure: Number; unit: participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants | 1 | 1
Statistical Analysis 1: Comparison: Monovalent Influenza Virus Vaccine vs Placebo; The percentage of subjects with fever was compared between the two treatment groups based on the upper limit of the two-sided 95% CIs for rate difference (monovalent vaccine minus placebo). The upper limit of the two-sided 95% CI was evaluated against the pre-specified equivalence criterion of 5 percentage points which corresponded to the following hypotheses: - H0 (null): rate difference ≥ 5 percentage points, - HA (alternative): rate difference < 5 percentage points; Test type: Non-Inferiority or Equivalence — Based on similar fever rate with 300 evaluable subjects (240 vaccine and 60 placebo recipients), the study would provide at least 98% power to rule out a rate increase of 5 percentage points assuming the true difference between the treatment groups is zero and the true fever rate is ≤ 1.0%. Power would be lower if the true difference was different from zero; score statistic; rate difference = -1.3, 95% CI 2-sided [-7.9 to 1.3]

2. Secondary Outcome: Number of Participants Reporting Any Solicited Symptom or at Least One Adverse Event (AE)
Description: Solicited symptoms were collected from administration of investigational product through Study Day 15. For this study, solicited symptoms included: fever (> 100°F oral), runny nose, sore throat, cough, vomiting, muscle aches, chills, decreased activity (tiredness), headache.
Time Frame: Days 1-8 after vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants
  Any solicited symptom | 97 | 23
  Fever > 100°F | 2 | 1
  Fever ≥ 101°F | 1 | 1
  Fever > 102°F | 0 | 0
  Fever > 103°F | 0 | 0
  Runny nose | 66 | 10
  Sore throat | 33 | 4
  Cough | 10 | 3
  Vomiting | 1 | 1
  Muscle aches | 15 | 4
  Chills | 0 | 0
  Decreased activity (tiredness) | 18 | 2
  Headache | 42 | 11
  Total participants reporting ≥ one AE | 27 | 2

3. Secondary Outcome: Number of Participants Reporting Any Solicited Symptom or at Least One AE
Time Frame: Days 1-15 after vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants
  Any solicited symptom | 102 | 25
  Fever > 100°F | 3 | 1
  Fever ≥ 101°F | 1 | 1
  Fever > 102°F | 0 | 0
  Fever > 103°F | 0 | 0
  Runny nose | 68 | 11
  Sore throat | 38 | 4
  Cough | 13 | 3
  Vomiting | 1 | 1
  Muscle aches | 16 | 4
  Chills | 1 | 0
  Decreased activity (tiredness) | 19 | 2
  Headache | 44 | 13
  Total participants reporting ≥ one AE | 29 | 3

4. Secondary Outcome: Number of Participants Reporting at Least One Serious Adverse Event (SAE) or New Onset Chronic Disease (NOCD)
Description: SAEs were those that resulted in death; were life-threatening; resulted in inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; were a congenital anomaly/birth defect in the offspring of a study participant; or were an important medical event that may have jeopardized the subject and may have required medical or surgical intervention to prevent one of the outcomes listed above. An NOCD was a newly diagnosed medical condition of a chronic, ongoing nature and assessed by the investigator as medically significant.
Time Frame: Days 1-29 after vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants
  Total participants reporting ≥ one SAE | 0 | 0
  Total participants reporting ≥ one NOCD | 0 | 0

5. Secondary Outcome: Number of Participants Reporting at Least One Serious Adverse Event (SAE) or New Onset Chronic Disease (NOCD)
Description: as for outcome 4
Time Frame: Days 1-181 after vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants
  Total participants reporting ≥ one SAE | 2 | 0
  Total participants reporting ≥ one NOCD | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time that written informed consent was obtained, AEs were collected through Day 15 after vaccination and SAEs were collected through Day 181 after vaccination.
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 2/240 | 0/60
Other Adverse Events (participants affected / at risk) | 23/240 | 3/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monovalent Influenza Virus Vaccine (N=240) | Placebo (N=60)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monovalent Influenza Virus Vaccine (N=240) | Placebo (N=60)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.